CLINICAL TRIAL: NCT00661570
Title: Amendment on Phase I Trial NO7VEG 'Assessment of a Next Generation Indwelling Provox Voice Rehabilitation System (Vega)
Brief Title: Long-term Clinical Feasibility of the New Indwelling Provox Vega 20 Voice Prosthesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary endpoint reached, slow accrual, leakage around
Sponsor: Atos Medical AB (Industry)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UD736
Record Dates: First submitted 2008-04-09; First posted 2008-04-18 (Estimated); Results first posted 2010-11-03 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Total Laryngectomy
Keywords: laryngectomy; larynx cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early feasability arm (Experimental)
  Interventions: Device: Provox Vega voice prosthesis (20 Fr)

INTERVENTIONS:
Device: Provox Vega voice prosthesis (20 Fr) — The current Provox2 voice prosthesis of laryngectomized patients will, when the patient comes in for a change, be replaced with a new, next generation Provox Vega voice prosthesis and insertion system
  Other Names: indwelling Provox voice prosthesis

SUMMARY:
The purpose of this study is to investigate long-term clinical feasibility of a new voice prosthesis and insertion system Provox Vega 20 with SmartInserter) for voice rehabilitation after total laryngectomy. Outcome measures are voice quality, ease of insertion, device life, and reason for replacement.

ELIGIBILITY:
Inclusion Criteria:

* total laryngectomy
* use Provox2 voice prosthesis
* at least two prior prosthesis changes

Exclusion Criteria:

* current puncture problems (f. ex. infection)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans JM Hilgers, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; Michiel WM van den Brekel, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the outpatient clinic when they came in for a voice prosthesis replacement.
Groups:
- Provox Vega 20: 26 Patients who normally use a Provox2 voice prosthesis, were asked to use a new Vega voice prosthesis with an outer diameter of 20 French.
Period: Overall Study
Arm/Group | Provox Vega 20
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Provox Vega 20
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.69 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Region of Enrollment [Number; unit: patients]
  Netherlands | 26

OUTCOME MEASURES:

1. Primary Outcome: Device Life Time
Description: Device life was measured from the time of insertion until the time of replacement. Reason for replacement was recorded. Only replacements for leakage through the device are considered for calculation of device life time.
Time Frame: at replacement of voice prosthesis (maximum 1 year)
Population: In 16 out of the 26 patients, the device was replaced for leakage through the device. These 16 devices were considered for calculation of device life time.
Measure: Median (Full Range); unit: days of use
Arm/Group | Provox Vega 20
Number analyzed (Participants) | 16
days of use | 93 (81.85) [3 to 279]

2. Secondary Outcome: Voice Quality
Description: Subjective patient opinion about 5 voice related items (intelligibility face to face and on the phone, loudness, pitch and fluency). The best value is 5 and the worst value is 20.
Time Frame: at 3 months or device change (whichever was first)
Population: 23 patients completed the structured questionnaires about the voice prosthesis. One patient received the wrong voice prosthesis after inclusion. Two patients had unsolvable leakage around the Provox Vega 20, which is 2.5 French smaller in outer diameter than their previous Provox2 voice prosthesis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Provox Vega 20
Number analyzed (Participants) | 23
Units on a scale | 8.4 (4.4)

3. Secondary Outcome: Ease of Insertion
Description: The Vega voice prosthesis used in this study is inserted with a new insertion tool, the SmartInserter. Physicians were asked to rate the insertion on a 4 point scale. what they thought of the new insertion tool, also in comparison to the regular tool used in the clinic, the Provox2 inserter. As the Provox voice prosthesis is a tool physicians already used, no insertions were performed with the Provox2 inserter during the study.
Time Frame: assessed immediately after insertion procedure
Population: All patients included for insertion evaluation
Measure: Number; unit: insertions
Arm/Group | Provox Vega 20
Number analyzed (Participants) | 26
insertions
  Not difficult at all | 20
  A little difficult | 4
  Rather difficult | 1
  Very difficult | 1

4. Secondary Outcome: Reason for Replacement
Time Frame: At removal of prosthesis
Population: 1 patient had his Vega inappropriately removed and received a Provox2.
Measure: Number; unit: patients
Arm/Group | Provox Vega 20
Number analyzed (Participants) | 25
patients
  leakage through prosthesis | 16
  periprosthetic leakage due to smaller diameter | 5
  combination of causes | 4

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time the new Vega prosthesis was inserted until the voice prosthesis was replaced.
Description: Adverse events were assessed after the insertion procedure, upon notification of a problem by the patient, and when the Provox Vega needed replacement. Normal reasons for replacement (leakage through, size changes) were not considered adverse events.
Arm/Group | Provox Vega 20
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No